CLINICAL TRIAL: NCT05014932
Title: Evaluation of Noise Induced by Ceramic-ceramic Friction Torques of Total Hip Prostheses With Customized Femoral Stem
Acronym: ATHENS
Status: Completed | Type: Observational
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-A02544-35
Record Dates: First submitted 2021-08-16; First posted 2021-08-20 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Arthroplasty Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Evaluation of noise induced by ceramic-ceramic friction torques of total hip prostheses with customized femoral stem.

Retrospective and prospective multicentric study.

DETAILED DESCRIPTION:
On a series of patients operated on for more than two years after a total hip arthroplasty that resulted in the implantation of a ceramic-on-ceramic prosthesis with a customized femoral stem:

Primary objective: To assess the frequency of occurrence of joint noise.

Secondary objectives:

* To describe the characteristics of the noise nuisance (date of onset, frequency, intensity, impact...)
* To evaluate the individual and surgical factors associated with the occurrence of noise pollution.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years or older, who has been informed of the research
* Patient who has had a fourth generation ceramic/ceramic hip replacement implanted for at least two years as a first-line replacement
* Patient who has had a three-dimensional preoperative examination leading to the design and implantation of a custom femoral stem
* Patient regularly monitored since surgery and for whom all clinical and radiological data are available at the three-month and two-year follow-up visits

Exclusion Criteria:

* Patient operated for revision
* Patient under legal protection, guardianship or curators
* Patient who has indicated his opposition to the use of his medical data (by completing and returning the non-opposition form which will be sent to him)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with at least two years of uncemented fourth generation ceramic/ceramic total hip replacement with customised femoral stem.
Sampling Method: Non-Probability Sample
Enrollment: 531 (Actual)
Dates: Start 2022-02-18 (Actual); Primary Completion 2023-03-14 (Actual); Study Completion 2023-03-14 (Actual)

PRIMARY OUTCOMES:
Noise nuisance | 2 years
  Percentage of occurrence of noise nuisance (assessed in relation to the total number of patients and the total number of prostheses).
  The frequency of occurrence of noise nuisance will be analysed descriptively. The time elapsed until the occurrence of the noise nuisance will be additionally assessed by a Kaplan-Meier analysis.

SECONDARY OUTCOMES:
Oxford Score | 2 years
  The Oxford Hip Score questionnaire (OHS 12) consists of 12 questions. It measures pain (6 items) and hip function (6 items) in relation to activities of daily living such as walking, dressing and sleep disturbance. Each question has 5 possible answers. Each has a value from 0 to 4, with 0 representing the highest level of severity and 4 representing no or almost no symptoms.
Hip disability and Osteoarthritis Outcome Score (HOOS) Score | 2 years
  The HOOS questionnaire is a self-administered questionnaire specific to hip arthroplasty. It consists of 40 questions with 5 domains: 5 questions on symptoms and stiffness; 10 questions on pain; 17 questions on functional results in daily life; 4 questions on sport and leisure activities; 4 questions on quality of life.
  It includes 5 sub-scores, one sub-score per domain.
Forgotten Joint Score | 2 years
  The Forgotten Joint Score (FJS-12) is a self-administered questionnaire consisting of 12 questions assessing the degree of forgetfulness of hip replacements in a given situation of daily life. Each answer is selected from a 5-point Likert scale with response options ranging from never (0) to most of the time (4).
Prosthesis life span | 2 years
  The life span of the prosthesis is the time between the implantation of the prosthesis and its complete or partial surgical revision.

CONTACTS AND LOCATIONS:
Overall Officials: Alexis NOGIER, MD PD, Principal Investigator — Clinique Maussins-Nollet
Locations (1):
- Clinique Maussins-Nollet, Paris, France